CLINICAL TRIAL: NCT04452292
Title: A Pilot Feasibility Study of Next Generation Sequencing-Based Stratification of Front Line Treatment of HighGrade Neuroendocrine Carcinoma
Brief Title: Next Generation Sequencing-Based Stratification of Front Line Treatment of HighGrade Neuroendocrine Carcinoma
Acronym: PRECISION-NEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Kunos (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor-Investigator, Charles Kunos, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20-GI-112-PMC; MULTI-37; KL2TR001996 (NIH); UL1TR001998 (NIH)
Record Dates: First submitted 2020-06-24; First posted 2020-06-30 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Large-Cell Neuroendocrine Carcinoma
Keywords: poorly differentiated neuroendocrine carcinoma; NGS; TP53/Rb1; co-mutation; molecular subtype
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No TP53/Rb1 Co-Mutation (Active Comparator): HG-LCNEC tumor lacking the TP53/Rb1 co-mutation (non-small cell-like).
  Interventions: Other: Treatment Specific for Non-Small Cell Carcinoma/Adenocarcinoma
- TP53/Rb1 Co-Mutation Present (Experimental): HG-LCNEC tumor with the TP53/Rb1 co-mutation.
  Interventions: Other: Treatment for Small Cell Lung Cancer

INTERVENTIONS:
Other: Treatment Specific for Non-Small Cell Carcinoma/Adenocarcinoma — Treatment assigned to targetable mutation. Or, for tumors that are by and large without any targetable mutation follow Large-Cell Neuroendocrine Carcinoma (NCCN) guideline-directed best front-line treatment for specific non-small cell carcinoma/adenocarcinoma.
  Arms: No TP53/Rb1 Co-Mutation
Other: Treatment for Small Cell Lung Cancer — Treatment assigned to a targetable mutation or the current standard-of-care regimen for the treatment of small cell lung cancer.
  Arms: TP53/Rb1 Co-Mutation Present

SUMMARY:
PRECISION-NEC is a single-center, open-label, pilot feasibility study of molecularly defined subtypes of metastatic high-grade neuroendocrine carcinoma (HG-NEC). The hypothesis is that HG-NEC (excluding small cell carcinoma) can be segregated based on mutational analysis and that next generation sequencing (NGS)-based assignment of therapy is feasible and will potentially improve the outcomes.

DETAILED DESCRIPTION:
Neuroendocrine tumors vary widely in both disease site and grade, ranging from low grade, relatively benign carcinoid tumors to aggressive and rapidly fatal high-grade neuroendocrine carcinomas. High-grade neuroendocrine carcinomas (HG-NECs) can originate anywhere in the body, and are highly aggressive, with dismal 5-year overall survival rates. The lung and gastrointestinal tract (small bowel, colon, rectum, or pancreas) form the majority of these HG-NECs sites. HG-NECs are classified into three subtypes based on histopathology, specifically, as small cell neuroendocrine carcinoma, large cell neuroendocrine carcinoma (LCNEC), or poorly differentiated neuroendocrine carcinoma.

There is a lack of consensus for upfront systemic regimens for HG-NECs and as such, treatment is often per physician preference. Most often, HG-NECs are treated with platinum-based chemotherapeutic regimens, with marked heterogeneity in response. It is well established that small cell neuroendocrine carcinomas are characterized by a co-mutation for TP53 and RB1, and are exceptionally platinum-sensitive. However less is known about LCNECs.

LCNEC was first introduced in 1991 by Travis et. al as a new type of lung cancer. The 2015 World Health Organization Classification categorized LCNEC under neuroendocrine tumors, along with typical carcinoma, atypical carcinoma and the more undifferentiated tumor represented by small cell lung cancer. Prior to 2015, LCNEC was classified under a general category of large cell carcinoma, however as pathologists studied this entity in detail, it was evident that LCNEC has a distinct clinicopathological identity. Histopathologically, these tumors are characterized by high mitotic rate (more than 10 mitosis per high power field), extensive necrosis, and neuroendocrine features, specifically the presence of chromogranin A, neuron specific enolase and synaptophysin.

LCNEC is a rare and aggressive disease with a paucity of data regarding disease progression. Precise incidence and prevalence is unknown. From 2003-2012, the Dutch Cancer Registry reported 952 histologically confirmed new cases of pulmonary LCNECs. Among these cases, 383 patients presented with advanced disease, primarily metastases to liver, bone, or brain. The prognosis is poor with overall 5-year survival for metastatic disease less than 5%, which is similar to small cell lung cancer (SCLC), although some studies suggest that the prognosis for early-stage LCNEC might be slightly better and similar to non-small cell lung cancer (NSCLC).

Molecular profiling of small-cell neuroendocrine carcinomas is well established and validated, indicating universally expressed co-mutation for TP53 and RB1. Recently there have been attempts to define genomic profiles of LCNEC. The development of a 241-gene panel on pulmonary tumors, next-generation sequencing allows LCNECs to be further defined.

Based on specific genetic signatures, Rekhtman and colleagues sub-classified 45 LCNECs into two major cohorts: 1) small cell-like (TP53/RB1 co-mutated; n=18) and 2) non-small cell-like (n=25), as well as one minor cohort (carcinoid-like n=2).

Similarly, molecular profiling of gastrointestinal high-grade neuroendocrine carcinomas (GI-NECs) indicate that they can also be dichotomously categorized by the presence or absence of co-mutations for TP53 and RB1.

Treatment regimens for small cell neuroendocrine carcinoma are well established, based on clinical trials conducted in SCLC. In contrast, current guidelines regarding optimal treatment for large-cell and poorly differentiated neuroendocrine carcinomas are nonexistent, driven by the paucity of data on these rare and highly fatal tumors. Additionally, the World Health Organization (WHO) recently defined a new subtype of high-grade neuroendocrine carcinoma, mixed neuroendocrine neoplasm (MINEN), which features characteristics found in large-cell carcinomas and in other tumor types, including adenocarcinomas for example.

To date, there are no prospective randomized clinical trials examining front line therapies for metastatic HG-NECs, based on mutational profiles. This study will utilize recent genomic profiles of high-grade large cell neuroendocrine carcinomas to guide and inform clinicians of optimal treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high grade neuroendocrine carcinoma that is metastatic and/or not resectable
* Adequate tissue available for genomic sequencing
* ECOG status less than or equal to 2
* Able to consent
* Patient received up to two cycles of chemotherapy prior to enrollment
* Adequate bone marrow function
* Adequate hepatic function
* Adequate renal function

Exclusion Criteria:

* Small cell carcinoma
* Psychiatric illness or social situations that limit compliance
* Pregnant and nursing women
* Patients who have completed more than two cycles of chemotherapy
* Patients with resectable cancer or eligible for curative therapy
* Patients with an actionable mutation for with guidelines recommend up-front therapy with targeted agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2023-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kunos, MD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saghaeiannejad Esfahani H, Vela CM, Chauhan A. Prevalence of TP-53/Rb-1 Co-Mutation in Large Cell Neuroendocrine Carcinoma. Front Oncol. 2021 May 31;11:653153. doi: 10.3389/fonc.2021.653153. eCollection 2021. PMID 34141612

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Opened to accrual in 11/2020 was closed to enrollment on 11/2022 due to poor accrual. Target accrual was 15 participants.
Period: Overall Study
Arm/Group | No TP53/Rb1 Co-Mutation | TP53/Rb1 Co-Mutation Present
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Closed to slow accrual and no participants were enrolled in TP53/Rb1 Co-Mutation Present arm
Groups:
- Total: Total of all reporting groups
Arm/Group | No TP53/Rb1 Co-Mutation | TP53/Rb1 Co-Mutation Present | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Sequencing Rate (Feasibility)
Description: Percentage of patients able to be sequenced within 2 months of the initial medical oncology visit.
Time Frame: 2 months
Population: Two participants were enrolled in this study. Due to the possibility that participants could reasonably be identified due to low enrollment, data cannot be presented.
Arm/Group | No TP53/Rb1 Co-Mutation | TP53/Rb1 Co-Mutation Present
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Molecular Cohort Assignment (Feasibility)
Description: Percentage of patients who were successfully assigned into a molecularly-defined cohort (TP53/RB1 co-mutations or not).
Time Frame: 2 months
Population: as for outcome 1
Arm/Group | No TP53/Rb1 Co-Mutation | TP53/Rb1 Co-Mutation Present
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Duration of time from the first cycle of anticancer therapy to time of progressive disease or death from any cause, whichever occurs first.
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | No TP53/Rb1 Co-Mutation | TP53/Rb1 Co-Mutation Present
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Complete Response Rate
Description: Percentage of patients experiencing overall complete response (CR).
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | No TP53/Rb1 Co-Mutation | TP53/Rb1 Co-Mutation Present
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Partial Response Rate
Description: Percentage of patients experiencing overall partial response (PR).
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | No TP53/Rb1 Co-Mutation | TP53/Rb1 Co-Mutation Present
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Progressive Disease Rate
Description: Percentage of patients experiencing overall progressive disease (PD).
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | No TP53/Rb1 Co-Mutation | TP53/Rb1 Co-Mutation Present
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Stable Disease Rate
Description: Percentage of patients experiencing overall stable disease (SD).
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | No TP53/Rb1 Co-Mutation | TP53/Rb1 Co-Mutation Present
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Only 2 participants were enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Description: Only 2 participants were enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | No TP53/Rb1 Co-Mutation | TP53/Rb1 Co-Mutation Present
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT04452292/Prot_SAP_ICF_000.pdf